CLINICAL TRIAL: NCT04927156
Title: Safety, Performance and Usability of BALT Medical Devices: The EVIDENCE Post Marketing Clinical Follow-up Platform. An International, Multicenter, Prospective, and Retrospective Data Collection
Brief Title: Safety, Performance and Usability of BALT Medical Devices: The EVIDENCE Post Marketing Clinical Follow-up Platform
Acronym: EVIDENCE
Status: Recruiting | Type: Observational
Sponsor: Balt Extrusion (Industry)
Responsible Party: Sponsor
Other Study IDs: CIP-202002-BALT DEVICES
Record Dates: First submitted 2021-06-09; First posted 2021-06-15 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Intracranial Aneurysm; Brain Arterial Disease; Acute Ischemic Stroke; Peripheral Vascular Diseases; AVM - Cerebral Arteriovenous Malformation; AVM; Fistulas Arteriovenous
Keywords: catheter; guidewire
MeSH Terms: conditions — Intracranial Aneurysm; Intracranial Arterial Diseases; Ischemic Stroke; Peripheral Vascular Diseases; Intracranial Arteriovenous Malformations; Arteriovenous Fistula

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- BALT medical devices
  Interventions: Device: BALT medical devices

INTERVENTIONS:
Device: BALT medical devices — Includes, but is not limited to, the following:
  * Access devices
  * Aneurysm treatment devices
  * Ischemic Stroke and peripheral occlusive diseases treatment devices
  * Arterio-Venous Malformations/fistulas treatment devices

SUMMARY:
BALT has designed an electronic platform to continue collecting clinical data as part of the post-marketing clinical follow-up of its devices.

This platform is purely exploratory, without hierarchical order of the objectives and associated outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Provision of a signed, written and dated informed consent or non-opposition (where applicable)

Exclusion Criteria

* Device(s) used in multiple procedures (two, or more, pathologies treated during the same procedure)
* Contra-indications of each device as described in the instructions for use.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include the BALT medical devices under consideration used in their respective indications for use during interventions performed at the participating sites.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-07-12 (Actual); Primary Completion 2041-06 (Estimated); Study Completion 2041-10 (Estimated)

PRIMARY OUTCOMES:
Rate of occurrence of device-specific safety indicator(s). | From the procedure to 12 months post-procedure depending on the device family.
  Specific outcomes will be adapted accordingly for each device family since the intended use will vary according to the device families.
Rate of devices achieving its intended use. | From the procedure to 12 months post-procedure depending on the device family.
  Specific outcomes will be adapted accordingly for each device family since the intended use will vary according to the device families.
Rate of devices achieving its specific performance indicator(s). | From the procedure to 12 months post-procedure depending on the device family.
  Specific outcomes will be adapted accordingly for each device family since the intended use will vary according to the device families.
Rate of devices in each category of the usability scale (Likert-type scale) for each usability indicator | From the procedure to 12 months post-procedure depending on the device family.
  Qualitative measurement of usability for each usability indicator (i.e., good, well adapted, fairly adapted, bad). Specific outcomes will be adapted accordingly for each device family since the intended use will vary according to the device families.

CONTACTS AND LOCATIONS:
Locations (12):
- France (6):
  - CHU Angers, Angers
  - Chu Bordeaux, Bordeaux
  - CHU Grenoble Alpes, La Tronche
  - Hôpital Roger Salengro, Lille
  - Kremlin Bicêtre - APHP, Paris
  - Chu Tours, Tours
- Halle, Halle, Germany
- Spain (5):
  - Hospital: Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico Universitario San Carlos, Madrid
  - Unversitario Central de Asturias, Oviedo
  - Hospital Universitario Marqués de Valdecilla (HUMV), Santander
  - Hospital Universitario Miguel Servet, Zaragoza

REFERENCES:
- See also: HDH — https://www.health-data-hub.fr/projets/securite-performance-et-utilisabilite-des-dispositifs-medicaux-balt-plateforme-de-suivi